CLINICAL TRIAL: NCT07328854
Title: 40.2Gy Versus 49.2Gy Radiotherapy in Low-Risk Target Volume for Chemosensitive Stage II Nasopharyngeal Carcinoma Under Full-Course Immunotherapy: a Multicentre, Randomised, Phase 3 Trial
Brief Title: 40.2Gy Versus 49.2Gy Radiotherapy in Low-Risk Target Volume for Chemosensitive Stage II Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.046
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Reduced-dose radiotherapy; Complete response; Partial response; Epstein-Barr Virus DNA; Low-risk target volume
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-dose radiotherapy to CTV2 combined with full-course immunotherapy (Experimental)
  Interventions: Drug: Cisplatin-based induction chemotherapy; Drug: Full course of PD-1 monoclonal antibody; Radiation: Reduced-dose radiotherapy to CTV2
- Conventional-dose radiotherapy to CTV2 combined with full-course immunotherapy (Active Comparator)
  Interventions: Drug: Cisplatin-based induction chemotherapy; Drug: Full course of PD-1 monoclonal antibody; Radiation: Conventional-dose radiotherapy to CTV2

INTERVENTIONS:
Drug: Cisplatin-based induction chemotherapy — Gemcitabine + cisplatin: Gemcitabine, 1,000 mg/m², Q3W, d1+d8, IV drip; cisplatin, 80 mg/m², Q3W, d1-3, IV drip. A total of 3 cycles.
  (Note: Gemcitabine can be replaced by docetaxel, albumin-bound paclitaxel, paclitaxel, etc.)
Drug: Full course of PD-1 monoclonal antibody — Tislelizumab 200 mg , once every 3 weeks (Q3W), intravenous infusion (iv). A total of 12 courses of treatment will be administered, including 3 courses during the induction chemotherapy phase, 3 courses during the radiotherapy phase, and 6 courses during the post-radiotherapy maintenance phase. Administration will start on Day 1 of induction chemotherapy and continue after the end of radiotherapy until the occurrence of intolerable toxicities, disease progression, withdrawal of consent, determination by the investigator that the patient needs to withdraw from treatment, or the completion of 12 courses, whichever comes first.
Radiation: Reduced-dose radiotherapy to CTV2 — GTV, 63.6Gy/30Fr/2.12Gy; CTV1, 54Gy/30Fr/1.8Gy; CTV2, 40.2Gy/30F/1.34Gy
  Arms: Reduced-dose radiotherapy to CTV2 combined with full-course immunotherapy
Radiation: Conventional-dose radiotherapy to CTV2 — GTV, 63.6Gy/30Fr/2.12Gy; CTV1, 54Gy/30Fr/1.8Gy; CTV2, 49.2Gy/30Fr/1.64Gy
  Arms: Conventional-dose radiotherapy to CTV2 combined with full-course immunotherapy

SUMMARY:
This study aims to explore the efficacy and adverse events of reduced-dose radiotherapy (40.2Gy) versus conventional-dose radiotherapy (49.2Gy) to low-risk target volume for chemosensitive intermediate-stage nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
This study intends to enroll low-risk intermediate-stage nasopharyngeal carcinoma patients who achieve CR/PR after induction chemotherapy and whose plasma EBV-DNA level has dropped to 0 or below the lower detection limit. These patients will be randomly assigned at a 1:1 ratio to receive either reduced-dose radiotherapy (40.2Gy) or conventional-dose radiotherapy (49.2Gy) to CTV2. Both groups will receive full-course immunotherapy. The study will follow up to observe differences in survival, adverse events, and quality of life between the two groups. It is expected that, on the premise of maintaining treatment efficacy, reducing the dose to CTV2 can decrease acute and chronic toxicities caused by radiotherapy and chemotherapy, thereby improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are informed of the basic content of this study and sign an informed consent form;
2. Age between 18 and 75 years;
3. Pathologically diagnosed as non-keratinising nasopharyngeal carcinoma (differentiated or undifferentiated, i.e., WHO type II or III);
4. Staged according to the 9th edition of the AJCC/UICC TNM classification as T1-3N2M0 or T3N0-1M0 (Stage II);
5. KPS ≥ 70;
6. Normal bone marrow function: WBC ≥ 4 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 90 g/L;
7. Imaging evaluation of treatment response after three cycles of GPP/TPP induction chemotherapy plus immunotherapy: CR or PR;
8. Plasma EBV DNA level decreases to 0 copies/mL or below the detection limit after induction chemotherapy;
9. Normal liver and kidney function: total bilirubin, AST, ALT ≤ 2.0 times the upper limit of normal, creatinine clearance ≥ 60 mL/min or creatinine ≤ 1.5 times the upper limit of normal.

Exclusion Criteria:

1. Patients with recurrent/metastatic nasopharyngeal carcinoma;
2. Pregnant or breastfeeding women (pregnancy tests should be considered for women of childbearing age; effective contraception should be emphasised during treatment);
3. Patients with a history of malignant tumours, excluding those who have undergone curative treatment for cervical cancer, basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer, or ductal carcinoma in situ;
4. Patients whose local/regional lesions have undergone radiotherapy or surgery (excluding diagnostic surgery), or whose lesions exhibit significant necrosis, making radiotherapy unsuitable or potentially leading to radiotherapy resistance;
5. Patients with other severe medical conditions that may pose significant risks or impair trial compliance. Examples include unstable cardiac disease requiring treatment, renal disease, hepatic disease, uncontrolled diabetes (fasting blood glucose > 1.5 × ULN), severe psychiatric disorders, or other malignant tumours;
6. Patients with a history of severe hypersensitivity reactions to any component of PD-1 monoclonal antibodies;
7. History of allergic reactions to the chemotherapy drugs used in this study (gemcitabine, docetaxel, albumin-bound paclitaxel, paclitaxel, cisplatin);
8. Patients with comorbidities requiring long-term use of immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive effects;
9. Patients with active tuberculosis, or those currently receiving antituberculosis treatment or who have received antituberculosis treatment within the past year prior to screening;
10. Other patients deemed ineligible for inclusion by the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.
Incidence of ≥3 grade adverse events | 3 years
  According to NCI-CTCAE 5.0, the proportion of patients who experienced ≥3 grade adverse events during treatment and follow-up.

SECONDARY OUTCOMES:
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomization to the date of first distant metastases.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Objective Response Rate (ORR) | 3 months
  Defined as the proportion of patients with tumor reduction achieving complete response (CR) or partial response (PR), assessed at 3 months after the end of concurrent chemoradiotherapy.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (15):
- China (15):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University cancer center, Guangzhou, Guangdong
  - the Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Central South University Cancer Hospital,, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang